CLINICAL TRIAL: NCT03345069
Title: Early Prediction of Cognitive and Motor Deficits Using Advanced MRI in Very Preterm Infants
Brief Title: Cincinnati Infant Neurodevelopment Early Prediction Study (CINEPS)
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other); Good Samaritan Hospital, Ohio (Other); Kettering Health Network (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: CIN_EARLYPREDICTION_001; 5R01NS094200 (NIH); 5R01NS096037 (NIH)
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Premature Infant
Keywords: Premature; Magnetic resonance imaging (MRI); Neurodevelopmental impairment; Cerebral Palsy; Cognitive Impairment; Diffusion MRI; Functional MRI; Infant; Magnetic resonance spectroscopy
MeSH Terms: conditions — Premature Birth; Cerebral Palsy; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants born very preterm: This is a single group prospective longitudinal, multisite cohort study of very preterm infants born at or below 32 weeks gestational age at birth

SUMMARY:
The Early Prediction Study is a longitudinal population-based cohort study for very preterm infants ≤32 weeks gestational age. Preterm infants recruited from three greater Cincinnati and two Dayton area neonatal intensive care units (NICUs) will undergo advanced MRIs at 41 weeks postmenstrual age and neurodevelopmental testing at the corrected ages of two and three years correct age. The goal of the Early Prediction Study is to accurately predict motor, cognitive, and behavioral deficits in individual very preterm infants using neuroimaging technologies and established epidemiologic approaches.

DETAILED DESCRIPTION:
With every neonatal intensive care unit discharge, physicians and early intervention specialists face a critical challenge: How to counsel parents about their very preterm infant's risk of developing cognitive and motor deficits and accurately assign early intervention therapies. More than 100,000 babies are born very preterm at ≤32 weeks gestational age every year in the United States. Up to 35% of these preterm survivors develop cognitive deficits, and up to 20% develop motor impairment. This places them at high risk for poor educational, health, and social outcomes. Yet reliable diagnosis of cognitive and motor deficits cannot be made until early childhood. This long and unnecessary delay wastes early intervention resources, dilutes the effectiveness of infant stimulation programs, and disrupts parental adaptation. Attempts to address these gaps with conventional neuroimaging and other approaches have failed. Thus, a critical need exists before neonatal discharge, to accurately predict cognitive and motor deficits in individual very preterm infants with the use of novel neuroimaging technologies and established epidemiologic approaches.

The investigators long-term research goal is to elucidate the etiology, pathogenesis, and early prediction of cognitive and motor deficits in order to facilitate preventive early interventions in very preterm infants, resulting in better outcomes. The investigators objectives in this application therefore are to:

1. Identify the clinical antecedents of objectively diagnosed diffuse white matter abnormality (DWMA).
2. Associate DWMA with pathologic changes on neuroimaging.
3. Predict cognitive and behavioral deficits at 3 years of age using objectively diagnosed DWMA in a geographic cohort of very preterm infants.
4. To predict motor impairment, especially cerebral palsy at 24 months corrected age.

The investigators central hypothesis is that objectively quantified DWMA is pathologic, associated with inflammation-associated perinatal illnesses, and an independent predictor of cognitive deficits at 3 years corrected age in very preterm infants. The investigators rationale for this research is that new knowledge investigators expect to have generated will enhance parental counseling, facilitate accurate risk stratification for early intervention therapies, and guide biologically-based strategies for early prevention of DWMA and cognitive and motor deficits in very preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized infants born at ≤32 weeks completed gestational age that are being cared for in all three level III/IV NICUs from the Greater Cincinnati area.

Exclusion Criteria:

* Infants with known chromosomal or congenital anomalies affecting the central nervous system or with cyanotic heart disease.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All very preterm infants (≤32 weeks completed gestational age) from a geographically-based population cared for in level III/IV NICUs in Cincinnati/Dayton are eligible. Those with known chromosomal or congenital anomalies affecting the central nervous system or with cyanotic heart disease will be excluded.
Sampling Method: Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Motor development | 2 years of age, corrected for prematurity
  Standardized assessment and diagnosis of cerebral palsy at 2 years corrected age
Cognitive development | 3 years of age, corrected for prematurity
  General Conceptual Ability (GCA) score from the Differential Abilities Scale, 2nd Edition
Behavioral development | 3 years of age, corrected for prematurity
  Scores on the Child Behavior Checklist & Early Childhood Behavior Questionnaire - Short Form

SECONDARY OUTCOMES:
Cognitive and language deficits at 2years of age | 2 years of age, corrected for prematurity
  Cognitive and language scores on Bayley Scales of Infant and Toddler Development, 3rd Ed
Executive function | 3 years of age, corrected for prematurity
  Computerized measures of executive function for preschoolers
Behavioral development | 3 years of age, corrected for prematurity
  General Adaptive Composite score on the Adaptive Behavior Assessment System, 2nd Ed.
Pre-academic skills | 3 years of age, corrected for prematurity
  Bracken School Readiness Assessment, 3rd Ed.

CONTACTS AND LOCATIONS:
Overall Officials: Nehal A Parikh, DO, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parikh NA. Advanced neuroimaging and its role in predicting neurodevelopmental outcomes in very preterm infants. Semin Perinatol. 2016 Dec;40(8):530-541. doi: 10.1053/j.semperi.2016.09.005. Epub 2016 Nov 15. PMID 27863706
- [Background] He L, Li H, Wang J, Chen M, Gozdas E, Dillman JR, Parikh NA. A multi-task, multi-stage deep transfer learning model for early prediction of neurodevelopment in very preterm infants. Sci Rep. 2020 Sep 15;10(1):15072. doi: 10.1038/s41598-020-71914-x. PMID 32934282
- [Result] Tamm L, Patel M, Peugh J, Kline-Fath BM, Parikh NA; Cincinnati Infant Neurodevelopment Early Prediction Study (CINEPS) Group. Early brain abnormalities in infants born very preterm predict under-reactive temperament. Early Hum Dev. 2020 May;144:104985. doi: 10.1016/j.earlhumdev.2020.104985. Epub 2020 Mar 9. PMID 32163848
- [Result] Parikh NA, Sharma P, He L, Li H, Altaye M, Priyanka Illapani VS; Cincinnati Infant Neurodevelopment Early Prediction Study (CINEPS) Investigators. Perinatal Risk and Protective Factors in the Development of Diffuse White Matter Abnormality on Term-Equivalent Age Magnetic Resonance Imaging in Infants Born Very Preterm. J Pediatr. 2021 Jun;233:58-65.e3. doi: 10.1016/j.jpeds.2020.11.058. Epub 2020 Nov 28. PMID 33259857
- [Result] Chandwani R, Kline JE, Harpster K, Tkach J, Parikh NA; Cincinnati Infant Neurodevelopment Early Prediction Study (CINEPS) Group. Early micro- and macrostructure of sensorimotor tracts and development of cerebral palsy in high risk infants. Hum Brain Mapp. 2021 Oct 1;42(14):4708-4721. doi: 10.1002/hbm.25579. Epub 2021 Jul 29. PMID 34322949
- [Result] Chen M, Li H, Fan H, Dillman JR, Wang H, Altaye M, Zhang B, Parikh NA, He L. ConCeptCNN: A novel multi-filter convolutional neural network for the prediction of neurodevelopmental disorders using brain connectome. Med Phys. 2022 May;49(5):3171-3184. doi: 10.1002/mp.15545. Epub 2022 Mar 14. PMID 35246986
- [Result] Lal SK, Nath LS. An atypical case of Vogt-Koyanagi syndrome. J Indian Med Assoc. 1986 Dec;84(12):382-3. No abstract available. PMID 3585016
- [Result] Jain VG, Kline JE, He L, Kline-Fath BM, Altaye M, Muglia LJ, DeFranco EA, Ambalavanan N, Parikh NA; Cincinnati Infant Neurodevelopment Early Prediction Study Investigators. Acute histologic chorioamnionitis independently and directly increases the risk for brain abnormalities seen on magnetic resonance imaging in very preterm infants. Am J Obstet Gynecol. 2022 Oct;227(4):623.e1-623.e13. doi: 10.1016/j.ajog.2022.05.042. Epub 2022 May 26. PMID 35644247
- [Result] Kline JE, Yuan W, Harpster K, Altaye M, Parikh NA. Association between brain structural network efficiency at term-equivalent age and early development of cerebral palsy in very preterm infants. Neuroimage. 2021 Dec 15;245:118688. doi: 10.1016/j.neuroimage.2021.118688. Epub 2021 Nov 7. PMID 34758381
- [Result] He L, Li H, Chen M, Wang J, Altaye M, Dillman JR, Parikh NA. Deep Multimodal Learning From MRI and Clinical Data for Early Prediction of Neurodevelopmental Deficits in Very Preterm Infants. Front Neurosci. 2021 Oct 5;15:753033. doi: 10.3389/fnins.2021.753033. eCollection 2021. PMID 34675773
- [Result] Chandwani R, Harpster K, Kline JE, Mehta V, Wang H, Merhar SL, Schwartz TL, Parikh NA. Brain microstructural antecedents of visual difficulties in infants born very preterm. Neuroimage Clin. 2022;34:102987. doi: 10.1016/j.nicl.2022.102987. Epub 2022 Mar 9. PMID 35290855
- [Result] Kline JE, Illapani VSP, Li H, He L, Yuan W, Parikh NA. Diffuse white matter abnormality in very preterm infants at term reflects reduced brain network efficiency. Neuroimage Clin. 2021;31:102739. doi: 10.1016/j.nicl.2021.102739. Epub 2021 Jun 25. PMID 34237685
- [Result] Li H, Chen M, Wang J, Illapani VSP, Parikh NA, He L. Automatic Segmentation of Diffuse White Matter Abnormality on T2-weighted Brain MR Images Using Deep Learning in Very Preterm Infants. Radiol Artif Intell. 2021 Feb 3;3(3):e200166. doi: 10.1148/ryai.2021200166. eCollection 2021 May. PMID 34142089
- [Result] Yuan W, Tamm L, Harpster K, Altaye M, Illapani VSP, Parikh NA. Effects of intraventricular hemorrhage on white matter microstructural changes at term and early developmental outcomes in infants born very preterm. Neuroradiology. 2021 Sep;63(9):1549-1561. doi: 10.1007/s00234-021-02708-9. Epub 2021 Apr 8. PMID 33830309
- [Result] Harpster K, Merhar S, Priyanka Illapani VS, Peyton C, Kline-Fath B, Parikh NA. Associations Between Early Structural Magnetic Resonance Imaging, Hammersmith Infant Neurological Examination, and General Movements Assessment in Infants Born Very Preterm. J Pediatr. 2021 May;232:80-86.e2. doi: 10.1016/j.jpeds.2020.12.056. Epub 2021 Jan 13. PMID 33453201
- See also: Early Prediction Study website — https://www.cincinnatichildrens.org/research/divisions/n/neonatology/labs/parikh/early-prediction-study